CLINICAL TRIAL: NCT01956539
Title: FREnch Survey on Heart Failure
Acronym: FRESH
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 12 680
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Observational Study
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: All patients over 18 years with chronic heart failure, and all patients hospitalized for acute heart failure de novo or not. The diagnosis of heart failure is the responsibility of the cardiologist including patient.

SUMMARY:
Heart failure is the most common heart disease with increasing incidence due to the aging of the population is improving the initial prognosis of various conditions that lead to more or less progressive heart failure.

Heart failure is of great variety of clinical and pathophysiological forms necessitating the creation of quality records to clarify each of these forms.

Many types of cardiomyopathies exist, some of which are infrequent but with specific care.

At the French level, few data exist. In addition, the therapeutic management changes regularly.

New European recommendations (endorsed by the French Society of Cardiology = FSC) were published in May 2012. Many therapeutic approaches are being evaluated. The course of care and how to take non-drug load (network monitoring, rehabilitation ...) have become important issues that have hardly been analyzed by existing records.

This also leads to better define the different forms of this disease, their natural history and methods of management applied in real life. The register of FSC follows the registry of the European Society of Cardiology (ESC)"Heart Failure (HF) Long Term" (CCTIRS No. 11.355bis) with inclusions will be completed in November 2012. This new study aims to generate more accurate data on a number of points and be more representative for a wider selection of patients, the French level.

DETAILED DESCRIPTION:
The recruitment period will be 24 months, with a day of inclusion for each week, which will be included both patients external consultant for chronic heart failure patients hospitalized in the cardiology department, during this day for acute heart failure.

Monitoring will be carried out 12 months during a consultation normally scheduled for this type of pathology with the cardiologist investigator. Patients included in a decompensation will also follow up to 3 months

ELIGIBILITY:
Inclusion Criteria:

* patient with chronic HF OR patient hospitalized foor acute HF de novo or not
* patient who accept to participate by signing a informed consent

Exclusion Criteria:

* patient who deny to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years with chronic heart failure, and all patients hospitalized for acute heart failure de novo or not. The diagnosis of heart failure is the responsibility of the cardiologist including patient.
Sampling Method: Non-Probability Sample
Enrollment: 2719 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Mortality at one-year of follow-up | 12 months
  Death rate at 12 months of follow-up

SECONDARY OUTCOMES:
Morbidity at one year of follow-up | 12 months
  Collect Chronic obstructive pulmonary disease (COPD) and diabetes mellitus during one year of follow-up, which frequently are associated with heart failure and impact patient outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lariboisiere, Paris, France

REFERENCES:
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the diagnosis and treatment of acute and chronic heart failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur J Heart Fail. 2008 Oct;10(10):933-89. doi: 10.1016/j.ejheart.2008.08.005. Epub 2008 Sep 16. No abstract available. PMID 18826876
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW; American College of Cardiology Foundation; American Heart Association. 2009 Focused update incorporated into the ACC/AHA 2005 Guidelines for the Diagnosis and Management of Heart Failure in Adults A Report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines Developed in Collaboration With the International Society for Heart and Lung Transplantation. J Am Coll Cardiol. 2009 Apr 14;53(15):e1-e90. doi: 10.1016/j.jacc.2008.11.013. No abstract available. PMID 19358937
- [Background] Heart Failure Society of America; Lindenfeld J, Albert NM, Boehmer JP, Collins SP, Ezekowitz JA, Givertz MM, Katz SD, Klapholz M, Moser DK, Rogers JG, Starling RC, Stevenson WG, Tang WH, Teerlink JR, Walsh MN. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2010 Jun;16(6):e1-194. doi: 10.1016/j.cardfail.2010.04.004. PMID 20610207
- [Background] Gheorghiade M, Zannad F, Sopko G, Klein L, Pina IL, Konstam MA, Massie BM, Roland E, Targum S, Collins SP, Filippatos G, Tavazzi L; International Working Group on Acute Heart Failure Syndromes. Acute heart failure syndromes: current state and framework for future research. Circulation. 2005 Dec 20;112(25):3958-68. doi: 10.1161/CIRCULATIONAHA.105.590091. No abstract available. PMID 16365214
- [Background] Nieminen MS, Bohm M, Cowie MR, Drexler H, Filippatos GS, Jondeau G, Hasin Y, Lopez-Sendon J, Mebazaa A, Metra M, Rhodes A, Swedberg K, Priori SG, Garcia MA, Blanc JJ, Budaj A, Cowie MR, Dean V, Deckers J, Burgos EF, Lekakis J, Lindahl B, Mazzotta G, Morais J, Oto A, Smiseth OA, Garcia MA, Dickstein K, Albuquerque A, Conthe P, Crespo-Leiro M, Ferrari R, Follath F, Gavazzi A, Janssens U, Komajda M, Morais J, Moreno R, Singer M, Singh S, Tendera M, Thygesen K; ESC Committe for Practice Guideline (CPG). Executive summary of the guidelines on the diagnosis and treatment of acute heart failure: the Task Force on Acute Heart Failure of the European Society of Cardiology. Eur Heart J. 2005 Feb;26(4):384-416. doi: 10.1093/eurheartj/ehi044. Epub 2005 Jan 28. No abstract available. PMID 15681577
- [Background] Tavazzi L, Maggioni AP, Lucci D, Cacciatore G, Ansalone G, Oliva F, Porcu M; Italian survey on Acute Heart Failure Investigators. Nationwide survey on acute heart failure in cardiology ward services in Italy. Eur Heart J. 2006 May;27(10):1207-15. doi: 10.1093/eurheartj/ehi845. Epub 2006 Apr 7. PMID 16603579
- [Background] Ezekowitz JA, Hernandez AF, Starling RC, Yancy CW, Massie B, Hill JA, Krum H, Diaz R, Ponikowski P, Metra M, Howlett JG, Gennevois D, O'Connor CM, Califf RM, Fonarow GC. Standardizing care for acute decompensated heart failure in a large megatrial: the approach for the Acute Studies of Clinical Effectiveness of Nesiritide in Subjects with Decompensated Heart Failure (ASCEND-HF). Am Heart J. 2009 Feb;157(2):219-28. doi: 10.1016/j.ahj.2008.10.002. Epub 2008 Nov 28. PMID 19185628
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Gheorghiade M, Abraham WT, Albert NM, Greenberg BH, O'Connor CM, She L, Stough WG, Yancy CW, Young JB, Fonarow GC; OPTIMIZE-HF Investigators and Coordinators. Systolic blood pressure at admission, clinical characteristics, and outcomes in patients hospitalized with acute heart failure. JAMA. 2006 Nov 8;296(18):2217-26. doi: 10.1001/jama.296.18.2217. PMID 17090768
- [Background] Metra M, Ponikowski P, Dickstein K, McMurray JJ, Gavazzi A, Bergh CH, Fraser AG, Jaarsma T, Pitsis A, Mohacsi P, Bohm M, Anker S, Dargie H, Brutsaert D, Komajda M; Heart Failure Association of the European Society of Cardiology. Advanced chronic heart failure: A position statement from the Study Group on Advanced Heart Failure of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2007 Jun-Jul;9(6-7):684-94. doi: 10.1016/j.ejheart.2007.04.003. Epub 2007 May 3. PMID 17481947
- [Background] Albert NM, Fonarow GC, Yancy CW, Curtis AB, Stough WG, Gheorghiade M, Heywood JT, McBride M, Mehra MR, O'Connor CM, Reynolds D, Walsh MN. Influence of dedicated heart failure clinics on delivery of recommended therapies in outpatient cardiology practices: findings from the Registry to Improve the Use of Evidence-Based Heart Failure Therapies in the Outpatient Setting (IMPROVE HF). Am Heart J. 2010 Feb;159(2):238-44. doi: 10.1016/j.ahj.2009.11.022. PMID 20152222
- [Background] Fonarow GC, Albert NM, Curtis AB, Stough WG, Gheorghiade M, Heywood JT, McBride ML, Inge PJ, Mehra MR, O'Connor CM, Reynolds D, Walsh MN, Yancy CW. Improving evidence-based care for heart failure in outpatient cardiology practices: primary results of the Registry to Improve the Use of Evidence-Based Heart Failure Therapies in the Outpatient Setting (IMPROVE HF). Circulation. 2010 Aug 10;122(6):585-96. doi: 10.1161/CIRCULATIONAHA.109.934471. Epub 2010 Jul 26. PMID 20660805